CLINICAL TRIAL: NCT02107651
Title: Serious Adverse Events in Patients Treated With New Oral Anticoagulants Are Underreported
Brief Title: Reporting of Adverse Events in Patients Treated With New Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Thue Bisgaard, Professor, Hvidovre University Hospital
Other Study IDs: 01675-HVH-2012-010-999
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Bleeding as Complication to Anticoagulation Therapy
Keywords: Bleeding; Anticoagulation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NOAC: Patients admitted for GI bleeding while in treatment with NOAC

SUMMARY:
Serious adverse events in patients treated with new oral anticoagulants are underreported.

DETAILED DESCRIPTION:
The study investigates if serious adverse events in patients treated with NOAC are reported to the Health and Medicines Authority.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for GI bleeding while in treatment with NOAC

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for GI bleeding while in treatment with NOAC
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients admitted with adverse event reported to authorities | Within one year of admission

CONTACTS AND LOCATIONS:
Overall Officials: Bisgaard Thue, Ph.D, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital University of Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Bay-Nielsen M, Kampmann JP, Bisgaard T. Gastrointestinal bleedings during therapy with new oral anticoagulants are rarely reported. Dan Med J. 2014 Nov;61(11):A4952. PMID 25370961